CLINICAL TRIAL: NCT00230308
Title: Identification and Characterization of Novel Proteins and Genes in Head and Neck Cancer
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB-11402; R01DE027750 (NIH)
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At the time of biospy or surgery, a small amount of tumor tissue (approximately 1 cc) will be taken from the main tumor specimen and stored until analysis.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Through this study, we hope to learn more about the mechanisms, which may contribute to development and progression of head and neck cancer. The long-term goal of this study will be to develop new strategies and drugs for the diagnosis and treatment of head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing surgery at Stanford University for head and neck cancer.

Exclusion Criteria:

Non-Stanford patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgery at Stanford University for head and neck cancer.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2002-04-02 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John B Sunwoo, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States